CLINICAL TRIAL: NCT04915872
Title: Are Standard Dosing Regimens of Piperacillin-Tazobactam Suitable in Critically Ill Patients With Open Abdomen and Negative Pressure Wound Therapy? A Population Pharmacokinetic Study.
Acronym: PK-LAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/53
Record Dates: First submitted 2021-02-01; First posted 2021-06-07 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Laparotomy; Critical Illness; Piperacillin, Tazobactam Drug Combination
Keywords: Open Abdomen; Negative Pressure Therapy; Antibiotics; Piperacillin - Tazobactam; Pharmacokinetics
MeSH Terms: conditions — Critical Illness | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample Urinary sample Negative Pressure Therapy fluid sample Peritoneal sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant: Critically Ill Patients with Open Abdomen and Negative Pressure Wound Therapy
  Interventions: Procedure: Blood sampling (T0, inclusion); Procedure: other samplings (T1)

INTERVENTIONS:
Procedure: Blood sampling (T0, inclusion) — Blood sample (5 ml) at 30 minutes after the loading dose of 4g/0.5g over 30 minutes for therapeutic drug monitoring at peak concentration (Cmax)
Procedure: other samplings (T1) — - T1 : Day of the first surgical revision, under PTZ administered by continuous infusion : Blood sample (5 ml) for therapeutic drug monitoring at steady state concentration (Css).
  Urinary sample and collection of urinary volume between T0 and T1 (Urinary Clearance) NPT fluid sample and collection of NPT volume between T0 and T1 (Peritoneal Clearance) Peritoneal sampling for therapeutic drug monitoring at the site of infection (CPt)

SUMMARY:
For several years, open abdomen with temporary abdominal closure using Negative Pressure Therapy (OA/NPT) has become one of the leading strategies to treat or prevent intra-abdominal hypertension in critically ill surgical patients after a wide range of complex abdominal injuries and conditions.

According to current practice, piperacillin-tazobactam (PTZ) is widely used as part of empirical combined antibiotic therapy to treat severe abdominal infections in the critically ill patients. On the other hand, little is known about the impact of OA/NPT on antibiotics pharmacokinetics and pharmacodynamics (PK/PD) and the optimal dosing regimens in this population remain unclear.

As PTZ is a small hydrophilic molecule with a very low level of protein binding, invesitigators hypothesized that OA/NPT should lead to significant changes in volume of distribution (Vd) and/or drug clearance (CL

The main objective of this study was to assess the incidence of underdosing and the pharmacokinetics of piperacillin in critically ill patients with OA/NPT.

The secondary objective was to assess the appropriateness of recommended regimens for empirical minimum inhibitory concentration (MIC) coverage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Admitted in surgical ICU for a suspected length of stay > 3 days
* Receiving an antimicrobial therapy by PTZ
* For an intra-abdominal infection
* Under OA/NPT during antimicrobial therapy
* With urinary and arterial catheters

Exclusion Criteria:

* Severe renal failure (CLCR < 30 ml/min) without indication for continuous renal replacement therapy (CRRT)
* Known allergy to PTZ
* Patient's refusal for participation to the research
* Patient unable to consent (dementia or severe psychiatric disorders, people under legal protection, people deprived of their liberty...)
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically Ill Patients with Open Abdomen and Negative Pressure Wound Therapy
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Rate of piperacillin | T1 (Day of the first surgical revision, up to 72 hours after inclusion)
  The main outcome investigated in this study was the rate of piperacillin (PIP) underdosing, arbitrarily defined by at least one of three samples under 16 mg/L. This threshold represents the highest MIC for Pseudomonas as per the European Committee on Antimicrobial Susceptibility Testing (EUCAST).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No